CLINICAL TRIAL: NCT07108205
Title: Clinical Study for Spectral Precise Image (SPI) Algorithm
Brief Title: Image Quality Study of Spectral Precise Image CT 7700
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-300450
Record Dates: First submitted 2025-05-19; First posted 2025-08-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Head; Body; Cardiac
Keywords: CT; Tomography; Image Quality; Noise reduction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Raw data will be reconstructed with iDose4: Raw data of subjects included in the study, following anonymization, will be transferred to Philips for reconstruction, raw data will be reconstructed with iDose4
  Interventions: Device: Paired reading analysis
- Raw data will be reconstructed with Spectral Precise Image: Raw data of subjects included in the study, following anonymization, will be transferred to Philips for reconstruction, raw data will be reconstructed with Spectral Precise Image
  Interventions: Device: Paired reading analysis

INTERVENTIONS:
Device: Paired reading analysis — Paired side be side evaluation Each reader will assess- Image Quality (IQ) & Diagnostic Confidence Ratings will be recorded using a 5-point Likert scale

SUMMARY:
The goal of the study is to evaluate the Image Quality (IQ), and diagnostic confidence of Spectral Precise Image for CT 7700 Scanner as compared with iDose4 as a standard-of-care reference.

DETAILED DESCRIPTION:
Spectral Precise Image is a reconstruction technique where the system uses a trained deep learning neural network to produce an image that reduces noise while improving low contrast detectability and maintaining the appearance of traditional filtered back projection (FBP) images.

Spectral Precise Image in Spectral CT 7700 system supports both conventional and spectral reconstructions.

The study will use raw data of subjects that are over the age of 22 years and scanned by Philips Spectral CT.

Study raw data, following anonymization, will be transferred to Philips for reconstructions, both conventional and spectral images will be reconstructed with iDose4 and with Spectral Precise Image at 100% dose.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects scanned by Spectral CT (K203020) according to the department standard of care clinical protocols.

  * Subjects age > twenty-two (22) years

Exclusion Criteria:

* • Scans that the site radiologists have deemed as non-diagnostic image quality in the standard practice (e.g. patient movement)

  * Scans that are not completed due to technical difficulties

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from subjects that met ALL of the inclusion criteria and NONE of the exclusion criteria will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Image Quality (IQ) of Spectral Precise Image reconstructions non inferior to iDose conventional images | 1 day
  Primary Endpoint (Co-Primary endpoints):
  1. The Image Quality (IQ) and diagnostic confidence of Spectral Precise Image reconstructions is at least as good as (non-inferior to) iDose4 for conventional images.
Image Quality (IQ) of Spectral Precise Image reconstructions non-inferior to iDose4 for spectral images of MonoE (MonoE 70Kev for Cardiac and for Body/ MonoE 66KeV for Head). | 1 day
  Primary Endpoint (Co-Primary endpoints): 2. The Image Quality (IQ) and diagnostic confidence of Spectral Precise Image reconstructions is at least as good as (non-inferior to)-iDose4 for spectral images of MonoE (MonoE 70Kev for Cardiac and for Body/ MonoE 66KeV for Head).

SECONDARY OUTCOMES:
Evaluation of the differences in Image Quality (IQ) of Spectral Precise Image reconstructions versus iDose conventional images | 1 day
  1. To evaluate the difference in Image Quality (IQ) and diagnostic confidence between Spectral Precise Image reconstructions for spectral images of MonoE (MonoE 70Kev for Cardiac and for Body/ MonoE 66KeV for Head) and iDose4 for conventional images.
Evaluation of the success rate for Spectral Precise Image reconstruction | 1 day
  2. To evaluate the success rate (%) for Spectral Precise Image reconstructions
Evaluation of the interobserver agreement level for the Co-Primary endpoints | 1 day
  3. The interobserver agreement level for the Co-Primary endpoints is more than 0.8.
Evaluation of images artifacts visualization and preservation of important features | 1 day
  4. Evaluation of images artifacts visualization and preservation of important features and clinical impact on diagnostic ability.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Montefiore, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Einstein, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided